CLINICAL TRIAL: NCT01811069
Title: Effect of Body Positioning on Upper Airway Patency During Induction of Anesthesia in Obese Patients
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yandong Jiang, Dr., Massachusetts General Hospital
Other Study IDs: 2012p-002632
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Obese
Keywords: Obese patients; Upper airway patency
MeSH Terms: conditions — Obesity | interventions — Smart Glasses

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Head up — 30˚ reverse trendelenburg body position

SUMMARY:
Upper airway obstruction (UAO) during induction of general anesthesia is a frequently occurring complication. The mechanism of UAO during anesthesia shares many similarities with the upper airway obstruction observed during obstructive sleep apnea (OSA). Obesity is major risk factors for OSA and obese patients have a higher prevalence of UAO during anesthesia. The change of body position improved upper airway stability during sleep in patients with OSA.We hypothesis that the 30˚ reverse trendelenburg body position maintain airway patency in obese patients during general anesthesia.

DETAILED DESCRIPTION:
This is a prospective, observational study. Fifteen subjects with BMI limited in the range of 30 kg/m2 to 50 kg/m2, between 18-65 years of age meeting ASA physical status classification I-III requiring general anesthesia for elective surgery will be recruited from the main operating room of the Massachusetts General Hospital. We will start the recruiting process at least 12 hours ahead of the surgery at a pre-admission test area.

The PI/Co-I who approaches a potential subject who has expressed interest will not be the anesthesiologist providing anesthesia care for the subjects. In addition the PI/Co-I approaching the patient will reinforce that she or he does not have to participate and that the decision not to participate will not affect their care at anytime.

The Principal Investigator or Co-Investigator will participate in the informed consent process in operative holding area. Subjects to be recruited will be given a thorough review of the informed consent, as well as the study purpose and procedures, and its risks, discomforts, and potential benefits. When the subject is comfortable with and knowledgeable about the protocol, he or she will sign the consent form in the presence of the investigator. Investigator will also sign the informed consent form. All subjects will be given ample time to read the consent form and consider participating in the trial. Any complaint or problems related to our recruitment plan will report in real time to the IRB.

ELIGIBILITY:
Inclusion Criteria:

BMI limited in the range of 30 kg/ m2 to 50 kg/ m2, 18-65 years of age ASA physical status classification I-III Requiring general anesthesia for elective surgery -

Exclusion Criteria:

1. Patients with major cardiovascular disease, respiratory disease, cerebral vascular disease or American Society of Anesthesiologists physical status class IV or greater.
2. Abnormal vital signs on the day of admission for surgery [heart rate (HR, >100 bpm or < 40 bpm), blood pressure (BP, >180/100 mmHg or < 90/60 mmHg), room air transcutaneous oxyhemoglobin saturation (SPO2) < 96%] that are not correctable with his or her routine medication or commonly used pre-operative medication.
3. Having claustrophobia and not able to tolerate the mask.
4. Any person with an anticipated difficult airway or those with a history of difficult airway who requires a fiberoptic intubation while awake.
5. Gastric-esophageal reflex disease that is refractory to treatment or a full stomach.
6. The subject has been in bed for more than 24 hours.
7. Neurological symptoms associated with neck extension, a neurological deficit from a previous stroke or spinal cord injury, a recent stroke or transient ischemic attack (TIA) within 2 weeks.
8. Pregnant women and women less than one month post-partum. Ruling out pregnancy will be conducted by careful history and physical examination as performed routinely prior to surgery. If the history is believed to be unreliable, the patient will be excluded unless a pregnancy test is performed and the result of the test is negative.
9. Emergency cases and subjects who have not adhered to the ASA NPO (Nil Per Os) guidelines.

   -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifteen patients with BMI limited in the range of 30 kg/ m2 to 50 kg/ m2, between 18-65 years of age meeting ASA physical status classification I-III requiring general anesthesia for elective surgery
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
expired tidal volume | 5 minutes
  The ventilation will continue for 1 min in flat position and then, operating table will be changed to 30˚ reverse trendelenburg position and the ventilation will continue for 1 min. Then, operating table will leveled and the ventilation will continue for 1 min.

SECONDARY OUTCOMES:
Vte/Area under the Curve (AUC) of the pressure trace during mask ventilation | 5 minutes
  The area under the airway pressure curve (AUC) defined as the area from the baseline pressure to the peak pressure during inspiration was calculated for evaluating pressure applied during inspiration.The AUC is a reflection of the change in mean airway pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Yandong Jiang, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States